CLINICAL TRIAL: NCT04248179
Title: The Ultrasound-guided Multiple-injection Costotransverse Block for Mastectomy and Primary Reconstructive Surgery. A Double Blind, Randomised, Placebo Controlled Trial.
Brief Title: The Ultrasound-guided Multiple-injection Costotransverse Block for Mastectomy and Primary Reconstructive Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZUH-MICB-UMPR
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
Keywords: Postoperative Pain; Opioid Consumption; Ultrasound guided nerve block; Paravertebral Block by proxy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Preoperative Multiple-injection Costotransverse Block (MICB) with three injections of each 10ml of Ropivacaine 5mg/ml corresponding to 3 * 10ml * 5mg/ml Ropivacaine = 150mg Ropivacaine.
  Interventions: Drug: Ropivacaine injection; Drug: Sufentanil and PONV prophylaxis
- Placebo (Placebo Comparator): Preoperative Multiple-injection Costotransverse Block (MICB) with three injections of each 10ml of Sodium chloride 9mg/ml corresponding to 3 * 10ml * 9mg/ml Sodium chloride = 189mg Sodium chloride.
  Interventions: Drug: Saline 0.9%; Drug: Sufentanil and PONV prophylaxis

INTERVENTIONS:
Drug: Ropivacaine injection — Ropivacaine 5mg/ml
  Arms: Active
Drug: Saline 0.9% — Saline 0.9%
  Arms: Placebo
Drug: Sufentanil and PONV prophylaxis — 30 minutes prior to emergence 0.2 μg/kg total body weight Sufentanil IV and 1 gram of paracetamol IV (if 6hrs since preoperative medicine) and 4 mg ondansetron IV (PONV prophylaxis) will be administered.
  Other Names: For postoperative pain and PONV treatment in the PACU

SUMMARY:
The investigators have developed a novel ultrasound-guided nerve block indicated primarily for breast cancer surgery that mimic a thoracic paravertebral block (TPVB) - hitherto the internationally accepted regional anesthesia golden standard for anesthesia of the hemithorax - but hypothetically without the risks of adverse events associated with the TPVB (i.e. pneumothorax, risk of bleeding in the thoracic paravertebral space, random and unmanageable epidural spread etc.). The investigators have already tested the anatomical- and block execution hypothesis in a randomized cadaveric study, and the investigators now have anatomical proof of concept for the functionality of the block technique. The investigators have also conducted a small clinical pilot study with very promising results. The investigators wish to conduct a randomized, placebo controlled and double-blind study, comparing the effect of the ultrasound-guided multiple-injection costotransverse block (MICB) vs. placebo. The aim with this study is to investigate the efficacy of the MICB vs. placebo in patients undergoing unilateral mastectomy and primary reconstructive surgery due to breast cancer or ductal carcinoma in situ. The hypothesis is, that the unilateral MICB will significantly reduce the opioid consumption during the first 24 postoperative hours and significantly reduce the Numerical Rating Scale pain score (0-10) and opioid related side effects.

DETAILED DESCRIPTION:
Twelve women in Denmark are diagnosed with breast cancer every day. Breast cancer and ductal carcinoma in situ (DCIS) are the primary type of cancer/precursor to cancer in women, and one of the main treatment modalities is surgical intervention. DCIS is a non-invasive (pre-malignant) condition in the breast with proliferating cells with malignant characteristics; confined in situ by the basal lamina in the breast. International DCIS is considered as manifest breast cancer, but in Denmark DCIS is considered as a precursor to breast cancer.

Breast cancer and DCIS surgery includes many subtypes ranging from the minor lumpectomy to major surgery; e.g. mastectomy and reconstructive surgery with or without axillary clearance. All surgical subtypes at the Department of Plastic Surgery and Breast Surgery, Zealand University Hospital (ZUH) are performed under general anesthesia (GA) and implies a multimodal pain regimen with preoperative oral medication (Paracetamol 1g, Celecoxib (NSAIDs) 400mg, Gabapentin 600mg, Dexamethasone 8mg and Dextromethorphan 30mg). Standard GA is total intravenous anesthesia (TIVA) and consists of Remifentanil, Propofol (and Rocuronium for tracheal intubation if needed), and the anesthesiologists will administer IV Sufentanil (a synthetic long-lasting opioid) 0.3-0.5 microg/kg 20-30 minutes prior to emergence for the immediate postoperative pain treatment. The patients are given additional Sufentanil and/or morphine intravenously in the post anesthesia care unit (PACU), if necessary.

Depending of surgical subtype, the surgeons will sometimes inject local anesthetic (LA) during surgery. The anesthesiologists will infrequently (depending on the availability of technical skills on the day of surgery) perform ultrasound-guided (USG) nerve blocks (Pecs 1 (and or) 2 and serratus anterior blocks) in the anterolateral thoracic wall prior to surgery, but this is not an implemented standard treatment. It is sadly neither national nor European standard to use USG nerve blocks for perioperative pain management for breast cancer and DCIS surgery. Instead, the vast majority of surgical centers rely heavily on the use of various long-lasting opioids, despite the adverse events associated with these drugs. Only relatively few surgical centers in Europe have implemented TPVB or other USG nerve blocks in the anterior thoracic wall as standard treatment for perioperative pain management.

USG multiple-injection TPVB is considered the regional anesthesia golden standard for breast cancer and DCIS surgery and reduces both acute and chronic pain as well as postoperative opioid consumption.

To determine which surgical subtype would be the most relevant to investigate (define the quantity of the research problem) the research group at ZUH have conducted a thorough retrospective study (including 111 patients) regarding postoperative pain and 12- and 24-hrs opioid consumption concerning patients undergoing breast cancer and DCIS surgery during 2016-2017 at the Department of Plastic Surgery and Breast Surgery, ZUH. The electronic anesthesia files, PACU files and ward files were meticulously reviewed. Six surgical subgroups were reviewed and the UMPR surgery elicited high values on the numeric rating scale (NRS) and a substantial need for perioperative opioids. The survey revealed an overall accumulated morphine consumption in the first 24 postoperative hours of 86.1±60.1mg (mean ± SD) of oral morphine equivalents (OME) and a NRS in the PACU of 4.5±2.4 (mean ± SD) in UMPR patients - and this surgical subtype was selected as most relevant and feasible to investigate. This dosage should be evaluated in relation to the standardized multimodal regimen described above.

There is definitely room for improvement in regards to the current treatment of this patient group. For instance, sub-group analysis reveals that patients having only received our current USG blocks (+preoperative oral medication and GA) have an accumulated morphine consumption in the first 24 postoperative hours of 81±55.2mg (mean ± SD) of OME.

Indication for UMPR surgery is either breast cancer or DCIS. UMPR surgery can be performed in several stages (and with several techniques) involving multiple GA techniques. However, at ZUH one-stage UMPR surgery is common and is described in the following (multiple stage surgery is irrelevant for the study protocol).

Standard operating procedure for one-stage UMPR surgery often involves two surgeons; i.e. one breast surgeon performing the mastectomy and one plastic surgeon performing the subsequent reconstructive surgery.

The mastectomy is skin conserving with incision inferolateral to the breast tissue. The breast tissue is removed leaving a pocket. The area profound to the major pectoral muscle and superficial to the minor pectoral muscle is opened and prepared for a prothesis. Very common this prothesis is an expander-prothesis with a filling-chamber (for subsequent ambulant re-fillings). An expander-prothesis is either permanent or temporary. If permanent the filling-chamber is removed ambulant with LA, if temporary the prothesis is removed in toto under GA and replaced with a permanent prothesis. Two surgical drains are installed; one in the pocket between the major pectoral muscle and the skin and one between the major pectoral muscle and the minor pectoral muscle (beside the prothesis). The drains exit the skin in the lateral thoracic wall without an exact defined anatomical point but often it is in the front axillary line below the incision.

The UMPR patient is evaluated by the operating surgeon around 14 days after surgery where the pathology results are reviewed.

Side effects of the current anesthesiologic practice/treatment. The use of morphine (IV and oral) can cause severe side effects, including nausea and vomiting, bowl paralysis, urine retention, sleep disturbances and respiratory depression. These side effects can delay mobilization after surgery, increase the risk of complications and worst of all be fatal.

In addition to all the well-known adverse events associated with morphine and the synthetic opioid derivate, these drugs have several masked adverse events (e.g. immunomodulation, hormonal disturbing, delirium triggering, angiogenetic etc.). Despite numerous (retrospective) studies regarding these issues, it is not yet possible to definitively link morphine consumption to metastasis formation and subsequent cancer recurrence. However, the surgical stress during the surgical procedures possibly generates an advantageous environment for dissemination of tumor cells when these inevitably are released to the blood stream by surgery. Studies advocate that TPVB reduces the perioperative opioid consumption - an indication of reduced surgical stress and other studies indicate that TPVB might even decrease the metastasis and progression of breast cancer. Large prospective studies regarding breast cancer recurrence with TPVB (and thoracic epidurals) are still ongoing.

Chronic postoperative pain Chronic postoperative pain (CPP) is a significant and very common problem associated to breast cancer and DCIS surgery ranging between 20-65% in all patients. Moderate to severe pain is reported to be between 10-20%. The underlying etiology is multifactorial and not fully understood, but it is suggested that CPP is occurring from a perioperative sensitization of the central nervous system. Numerous studies suggest that TPVB might decrease CPP and it has been postulated that the effect is due to an efficient treatment of acute pain leading to a decreased sensitization (both peripheral and central sensory) and a lower incidence of CPP.

A new prospective observational study finds that severity of acute pain is associated with the development of persistent pain.

The new block. The breast is innervated by the lateral and medial pectoral nerves from the brachial plexus and the T2-T6 thoracic spinal nerves. Hence, no regional technique will block the entire hemithorax with a single injection. The relatively new USG nerve blocks in the anterior thoracic wall like the "pecs block" and serratus anterior plane block, do not target the same nerves as TPVB.

The TPVB is executed in the posterior thoracic wall near the vertebral bodies with the needle tip just adjacent to the pleura and thereby with an inherent risk of pneumothorax as well as other serious adverse events. In expert hands and with ultrasound guidance the risk is probably relatively low. However, many anesthesiologists are still reluctant to perform the block due to the perceived risks.

Recently, the erector spinae plane block (ESPB) emerged and quickly gained a lot of attention for various indications. The ESPB have only been used for breast cancer surgery in a few case studies and in one RCT but presumably with some success.

The investigators have modified the ESPB to a novel multiple-injection costotransverse block (MICB). MICB is also a USG nerve block in the posterior thoracic wall. With MICB, the investigators inject LA on the superficial side of the superior costotransverse ligament (SCTL); which is the posterior border of the thoracic paravertebral space (TPVS). The LA will spread from the injection point and into the TPVS via the costotransverse foramen and the veins traversing the SCTL. Thereby the investigators mimic a TPVB, but - very important - with the needle tip in a very comfortable distance to the pleura reducing the risk of adverse events. The investigators have already proved this in a large cadaveric study with multinational collaboration. In this study, the MICB effectively stained the ventral rami, the communicating rami and the thoracic sympathetic trunk. Epidural spread was completely absent with the MICB.

The investigators have published two abstracts concerning this new block modality - and the main article is published in Acta Anaesthesiologica Scandinavica.

Pilot studies show that the MICB is considered a PNB with very little discomfort for the patient (NRS 1-2) "as painful as having a standard IV line in the hand" - which aligns with a previous study performed in our department regarding a deep nerve block for analgesia of the abdominal wall.

As the end-point for the MICB is the analgesic effect of a TPVB the investigators find it relevant to describe the contraindications to TPVB.

In general, there are few contraindications to TPVB. However, infection at the site of needle insertion, empyema, allergy to local anesthetic drugs, patient refusal and tumor occupying the TPVS are the most common noted contraindications in the literature. Before the emergence of ultrasound for nerve block execution coagulopathy, bleeding disorder or therapeutic anticoagulation were considered as relative contraindications for TPVB. Today, with ultrasound guidance there are no firm consensus on relative contraindications regarding especially therapeutic anticoagulation when performing TPVB.

Every day the investigators perform deep truncal blocks at the department at ZUH and the investigators have yet to see bleeding as a complication. The MICB is NOT a neuraxial block, neither do the investigators consider it a deep block. The mere purpose of the MICB is to further reduce the already low incidence of complications with TPVB. Recently, one accidental pneumothorax (with TPVB) was reported in well over 2000 patients, but not a single bleeding complication was reported and another study with 1427 TPVBs only six complications was reported (no bleeding); all handled successfully.

The investigators generally consider the MICB (and other paravertebral blocks by proxy) as safe procedures.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective unilateral mastectomy and primary reconstructive (UMPR) surgery with subpectoral implant due to breast cancer and ductal carcinoma in situ
* Age 18 years or above at the date of inclusion
* Have received thorough information, orally and in written, and signed the "Informed Consent" form on participation in the study.

Exclusion Criteria:

* Scheduled for elective UMPR surgery due to breast cancer and DCIS combined with simultaneous contralateral major breast surgery* (mastectomy, mastopexy and subpectoral breast reconstruction). Minor contralateral surgery (e.g. lipofilling) are accepted.
* Scheduled free flap reconstructive surgery
* Inability to cooperate
* Inability to speak, read and understand Danish
* Allergy to local anaesthetics or opioids
* Daily intake of opioids, according to the investigators decision
* Illegal drug and/or substance abuse, according to the investigators decision
* Local infection at the site of injection or systemic infection
* Difficult sonoanatomical visualisation of the target area (SCTL, ITTC etc.) necessary for the block execution
* Substantial co-morbidity, ASA>3
* Severe hypovolemia
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Morphine Consumption | 24 hours
  The primary aim of this study is total morphine consumption in the first 24 postoperative hours (data from PCA pump and the patient's medical record).

SECONDARY OUTCOMES:
Pain intensity | 24 hours
  Pain intensity (NRS 0-10/10) in the study period at T0 (arrival in the PACU), after 15 minutes, 30 minutes, 45 minutes and one hour.
  And pain intensity (NRS 0-10/10) in the intervals
  * [ arrival at the ward - 4 hrs. postop ]
  * ] 4 hrs. postop - 8 hrs. postop ]
  * ] 8 hrs. postop - 12 hrs. postop ]
  * ] 12 hrs. postop - 16 hrs. postop ]
  * ] 16 hrs. postop - 20 hrs. postop ]
  * ] 20 hrs. postop - 24 hrs. postop ]
Morphine consumption at 4, 8, 12, 16 and 20 postoperative hours. | 20 hours
  NRS score will be recorded electronically in the PCA-pump when morphine is administrated. All patients must enter NRS 0-10 on the PCA pump prior to morphine bolus administration.
Duration of block (time to first opioid). | 24 hours
  How long time does the MICB work?
Patient satisfaction with application of the block. | Immediately after application
  Patient is asked immediately after block application, Numeric Rating Scale (0-10, 0 = no pain, 10 = worst pain)
The degree of morphine-related side effects (PONV, itching, fatigue, etc.). | 24 hours
  PONV. 0-3; 0=No nausea. 3=Unmanageable nausea
Time from operation (T0) to ambulation (bed to chair to walking) | 24 hours
  When is the patient capable to ambulate; ie. going to the bathroom by themself
Time to discharge (days). | 5 days (anticipated)
  When is the patient discharged?
Quality of recovery | 24 hours and 14 days
  Quality of Recovery - 15 score (QoR15). Preoperatively compared to twice postoperatively. Preoperatively the patients are asked to fill in the validated Quality of Recovery Questionnaire QoR1536 questionnaire repeated at T0+24hrs. and 14 days after surgery (possibly by phone interview). The QoR15 questionnaire results in a score of 0-150.

CONTACTS AND LOCATIONS:
Overall Officials: Jens N Børglum, PhD, MD, Study Director — Department of Anaesthesiology, Zealand University Hospital, Roskilde
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Zealand University Hospital, Roskilde, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nielsen MV, Moriggl B, Hoermann R, Nielsen TD, Bendtsen TF, Borglum J. Are single-injection erector spinae plane block and multiple-injection costotransverse block equivalent to thoracic paravertebral block? Acta Anaesthesiol Scand. 2019 Oct;63(9):1231-1238. doi: 10.1111/aas.13424. Epub 2019 Jul 23. PMID 31332775